CLINICAL TRIAL: NCT00432250
Title: The Use of Cervical Length to Reduce Hospital Stay in Women Admitted Because of Preterm Labor.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CLHSPTL
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2007-02-07 (Estimated); Status verified 2007-02

CONDITIONS: Labor, Premature; Cervical Length
Keywords: Preterm labor; Cervical ultrasonography; Hospital stay
MeSH Terms: conditions — Obstetric Labor, Premature

INTERVENTIONS:
Procedure: Cervical length ultrasound

SUMMARY:
The objective of this study was to investigate the effect of the use of sonographic cervical length (CL) on the hospital stay in women admitted because of preterm labor.

DETAILED DESCRIPTION:
Eligible women who agreed to participate in the study were randomized by means of a central randomization office into two groups:

CONTROL group: cervical length was measured but the result was blinded to the physician in charge and women was managed according to the standard protocol.

STUDY group: cervical length was measured and the result was reported to the physician in charge. If cervical length was of 25 mm or more, discharge in 12-24 h was recommended. If cervical length was less than 25 mm, decision on discharge was made following clinical criteria.

ELIGIBILITY:
Inclusion Criteria:

* Admitted because of preterm labor
* Not delivered after 24-48 h of admission
* Single pregnancy
* Intact membranes
* Gestational age between 24.0 and less tahn 36.0 weeks
* Bishop score < 6

Exclusion Criteria:

* Fetal death or malformation
* Signs of chorioamnionitis
* Non-reassuring fetal test

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-01; Study Completion 2005-04

PRIMARY OUTCOMES:
Length of hospital stay
Gestational age at delivery

SECONDARY OUTCOMES:
Rate of hospital stay below 3 days
Interval admission-to-delivery < 7 days
Rate of preterm delivery before 37 weeks
Rate of preterm delivery before 34 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Montse Palacio, Principal Investigator — Hospital Clinic of Barcelona; Vicenç Cararach, Principal Investigator — Hospital Clínic of Barcelona
Locations (1):
- Hospital Clínic of Barcelona, Sabino de Arana 1, Barcelona, Spain